CLINICAL TRIAL: NCT01605812
Title: Phase 1 Evaluate Capsular Apposition to Intraocular Lens in Subjects With High Myopia by Ultra-long Scan Depth Optical Coherence Tomography; Phase 2 Evaluate Capsular Apposition to Different Types of Intraocular Lens in Subjects
Brief Title: Evaluate Capsular Apposition to Intraocular Lens
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, doctor of ophthalmology, Principal Investigator, Clinical Professor, Wenzhou Medical University
Other Study IDs: WZYXY-ZYY-OCT
Record Dates: First submitted 2012-05-11; First posted 2012-05-25 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Capsule Opacification; Tissue Adhesions; Aphakia - Lens Capsule Present; Opacification of Intraocular Lens
Keywords: IOL;; capsule；; PCO;; OCT
MeSH Terms: conditions — Capsule Opacification; Tissue Adhesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- high myopia: high myopia (axial length>26mm)
- emmetropia: emmetropia (22<axial length<25mm) as control group.

SUMMARY:
In this study, the investigators examined the capsule-IOL interaction including anterior and posterior capsule adhesion, contact between posterior capsule and the posterior edge of intraocular lense (IOL), configuration of capsular bend and the incidence of posterior capsular opacity (PCO) between high myopia eyes and emmetropia eyes.

DETAILED DESCRIPTION:
150 eyes of 150 cataract patients scheduled for phacoemulsification surgery were recruited, of which 20 eyes were high myopia (AL > 26mm) and 40 eyes were emmetropia (22 < AL < 25mm) as control group.High myopia eyes and 20 emmetropia eyes were implanted with the single-piece hydrophobic acrylic IOL (Acrysof IQ SN60WF, Alcon laboratories, Inc. IQ group). Another 20 emmetropia eyes were implanted with the other single-piece hydrophilic acrylic IOL (Akreos Adapt, Bausch &Lomb, AO group).80 eyes implanted with the single-piece hydrophobic acrylic IOL were examined by SSOCT to build the 3-D model of anterior segment.

Methods: 60 eyes were examined by custom-built UL-OCT at 4 hours, 1 day, 7 day, 14 day, 28 day, 3 month, 6 month,12 month after surgery.30 eyes implanted with the single-piece hydrophobic acrylic IOL were recruited for evaluation of the SSOCT reliability.50 eyes were examined by SSOCT at 1 day, 7 day,1 month, 3 months,6 months,12 months after surgery.

Measures: Contact of the anterior and posterior lens capsule with the IOL optic surface was evaluated. Types of capsular bend were described at the last follow-up. The incidence of posterior capsular opacity (PCO) was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with an AL of 26.00mm or more were recruited to the high myopia group.
* Eyes with an AL of 22.00 to 25.00 mm were recruited to the emmetropia group.

Exclusion Criteria:

* Preoperative exclusion criteria included diabetes, history of ocular surgery or inflammation, pupils could not be dilated over 7mm after mydriasis,
* patients who could not be available for follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective study consisted consecutive patients with high axial myopia (myopia group) and age-matched patients with normal axial length (control group). All eyes underwent uncomplicated phacoemulsification with a single-piece IOL (AcrySof, Alcon) implantation for cataract treatment.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate Capsular Apposition to Intraocular Lens in high myopia eyes and emmetropia eyes with different types of IOL | 4hour, 1day, 7day, 14day, 28day, 3month, 6month, 12month

CONTACTS AND LOCATIONS:
Overall Officials: yune zhao, MS, Study Chair — Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Tao A, Lu P, Li J, Shao Y, Wang J, Shen M, Zhao Y, Lu F. High resolution OCT quantitative analysis of the space between the IOL and the posterior capsule during the early cataract postoperative period. Invest Ophthalmol Vis Sci. 2013 Oct 25;54(10):6991-7. doi: 10.1167/iovs.13-12849. PMID 24065808